CLINICAL TRIAL: NCT01781143
Title: Self-operated Endo-vaginal Telemonitoring (SOET), an Economic and Patient-empowered Method for Ovarian Stimulation for In-vitro Fertilization (IVF).
Acronym: SOET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Flanders Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011/669
Record Dates: First submitted 2013-01-21; First posted 2013-01-31 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: IVF Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perform echo at home. (Experimental): A group of women that follows an IVF treatment, will perform their echoes at home, instead of always make an appointment in the clinic.
  Interventions: Device: Perform Echo at home.

INTERVENTIONS:
Device: Perform Echo at home. — A group of women that follows an IVF treatment, will perform their echoes at home, instead of always make an appointment in the clinic.
  Other Names: A home echo system will be used to perform an echo.

SUMMARY:
The SOET project introduces a new strategy for routine follow-up of follicle growth during the hormonal treatment phase of an in-vitro fertilization (IVF) treatment cycle. After a learning instruction and demo, patients should be able to perform most of their vaginal echoes at home. The images can be sent to the medical center over the internet. These images are analyzed by the expert.

ELIGIBILITY:
Inclusion Criteria:

* Woman, suffering from subfertility.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Higher efficacy by taking an echo at home. | Every 2 days, up to a year.
  During an IVF treatment, women are asked to perform the echo themselves, at home. This should create higher efficacy: patients are less stressed and can choose the moment of taking the echo themselves. Furthermore, this should result in a more cost effective and time saving way.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gerris, Ph.D, M.D., Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (4):
  - University Hospital VUB, Brussels
  - Hospital Oost-Limburg, Genk
  - Ghent University Hospital, Ghent
  - Clinique Saint-Vincent, Rocourt

REFERENCES:
- [Derived] Gerris J, Delvigne A, Dhont N, Vandekerckhove F, Madoc B, Buyle M, Neyskens J, Deschepper E, De Bacquer D, Pil L, Annemans L, Verpoest W, De Sutter P. Self-operated endovaginal telemonitoring versus traditional monitoring of ovarian stimulation in assisted reproduction: an RCT. Hum Reprod. 2014 Sep;29(9):1941-8. doi: 10.1093/humrep/deu168. Epub 2014 Jul 3. PMID 24993931
- See also: Related Info — http://www.uzgent.be